CLINICAL TRIAL: NCT00444041
Title: Pre- and Postoperative Chemotherapy Including Bevacizumab in Potentially Curable Metastatic Colorectal Cancer (mCRC). A Multicenter, Single Arm Phase I/II Academic Trial
Brief Title: Pre- and Postoperative Chemotherapy Including Bevacizumab in Potentially Curable Metastatic Colorectal Cancer
Acronym: ASSO-LM1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austrian Society Of Surgical Oncology (Other)
Responsible Party: Principal Investigator, Univ.Prof.MD Thomas Grünberger, Prof, Austrian Society Of Surgical Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO-ASSO-LM1
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; surgery; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xelox, Bev (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — neoadjuvant therapy prior to elective surgery

SUMMARY:
Major attempt is being given to the potential of curing patients with metastatic colorectal cancer due to the recognition of dramatic change in survival figures achieved in palliative chemotherapy combination treatment protocols. Achieving resectablity rates in previously unresectable patients has been defined as study endpoint among other well known primary and secondary objectives. Curing metastatic colorectal cancer is most likely in resectable patients and therefore the logical next step after completion of chemotherapy combination studies (e.g. EORTC 40983) is the addition of targeted agents. Bevacizumab has the most valid data of improving outcome figures and was therefore chosen as additional agent. Safety of the combination with Xelox was demonstrated in the investigators pilot trial (Gruenberger JCO 2006, ASCO 2006, WCGC 2006, ESMO 2006), consequently response rate and resection rate will be the primary endpoints in this trial.

STUDY OBJECTIVES

Primary Objective The primary objective of this study is the Resectability (R0) rate after neoadjuvant Bevacizumab in potentially resectable mCRC.

Secondary Objectives The secondary objectives of this study include

* Feasibility with regards to GI bleeding and wound healing complications after surgery of liver metastases
* General safety
* Overall Response Rate (ORR)
* Recurrence Free Survival (RFS)
* Overall Survival (OS)

STUDY DURATION Recruitment is planned for 12 months. Patients will be treated for 6 cycles XELOX and 5 cycles Bevacizumab. Surgery will be performed 2 weeks after the last Capecitabine administration, allowing a time window of 5 weeks between the last Bevacizumab administration and surgery.

Therapy with 6 cycles of XELOX and Bevacizumab will be restarted 4-5 weeks after surgery.

With a Follow up period of 2 years after the last enrolled patient, in order to assess RFS and OS, the trial will last for approx. 3 years.

NUMBER OF CENTRES Four centres with a high level of experience in the surgery of liver metastases are planned to participate in this study.

SELECTION CRITERIA

Total Number of Patients and Target Population The planned total sample size for this study is 43 patients. Patients with potentially resectable metastatic colorectal cancer previously untreated for metastatic disease will be enrolled in this trial.

DETAILED DESCRIPTION:
Major attempt is being given to the potential of curing patients with metastatic colorectal cancer due to the recognition of dramatic change in survival figures achieved in palliative chemotherapy combination treatment protocols. Achieving resectablity rates in previously unresectable patients has been defined as study endpoint among other well known primary and secondary objectives. Curing metastatic colorectal cancer is most likely in resectable patients and therefore the logical next step after completion of chemotherapy combination studies (e.g. EORTC 40983) is the addition of targeted agents. Bevacizumab has the most valid data of improving outcome figures and was therefore chosen as additional agent. Safety of the combination with Xelox was demonstrated in our pilot trial (Gruenberger JCO 2006, ASCO 2006, WCGC 2006, ESMO 2006), consequently response rate and resection rate will be the primary endpoints in this trial.

STUDY OBJECTIVES

Primary Objective The primary objective of this study is the Resectability (R0) rate after neoadjuvant Bevacizumab in potentially resectable mCRC.

Secondary Objectives The secondary objectives of this study include

* Feasibility with regards to GI bleeding and wound healing complications after surgery of liver metastases
* General safety
* Overall Response Rate (ORR)
* Recurrence Free Survival (RFS)
* Overall Survival (OS)

STUDY DURATION Recruitment is planned for 12 months. Patients will be treated for 6 cycles XELOX and 5 cycles Bevacizumab. Surgery will be performed 2 weeks after the last Capecitabine administration, allowing a time window of 5 weeks between the last Bevacizumab administration and surgery.

Therapy with 6 cycles of XELOX and Bevacizumab will be restarted 4-5 weeks after surgery.

With a Follow up period of 2 years after the last enrolled patient, in order to assess RFS and OS, the trial will last for approx. 3 years.

NUMBER OF CENTRES Four centres with a high level of experience in the surgery of liver metastases are planned to participate in this study.

SELECTION CRITERIA

Total Number of Patients and Target Population The planned total sample size for this study is 40 patients. Patients with potentially resectable metastatic colorectal cancer previously untreated for metastatic disease will be enrolled in this trial.

STUDY DESIGN

Design This is a single arm, multicenter Phase I/II trial to evaluate the Resectability (R0) rate after neoadjuvant Bevacizumab in combination with a biweekly regime of capecitabine plus oxaliplatin (XELOX) in potentially resectable mCRC.

The pre-operative treatment phase consists of 6 cycles XELOX and 5 cycles Bevacizumab. The cycle duration is 2 weeks.

Surgery will be performed 2 weeks after the last administration of Capecitabine, allowing a time window of 5 weeks between the last dose of Bevacizumab and surgery.

The post-operative treatment phase consists of 6 cycles XELOX + Bevacizumab and will be re-started 4-5 weeks after surgery.

Patients will be further followed for tumour progression and survival for a further 2 years after the last patient has been enrolled in this trial (end of the study follow up).

Schedule of Assessment and Study Procedures Study assessments and procedures will be performed as shown in Table 1 and 2. Screening and Baseline Written informed consent must be obtained prior to the patient undergoing any study-specific procedures.

1. Tumor assessments: abdominal and pelvic CT / MRI and chest CT / MRI may be obtained up to 4 weeks prior to enrollment.
2. Assessments to be made up to 14 days before enrollment include: demographic data, medical history, cancer/treatment history, concomitant disease/treatment, physical examination (including basic neurologic exam by investigator), electrocardiogram (ECG) and CEA, CA 19-9 determination.
3. Assessments to be made within 7 days before enrollment: height, weight, vital signs (body temperature, blood pressure, and pulse/heart rate), ECOG Performance Status, hematology, blood chemistry (including creatinine clearance calculation), INR & aPTT, serum pregnancy test (for all women less than 2 years amenorrheic), dipstick urinalysis for proteinuria, and 24-hour urine collection for determination of total protein (if necessary).
4. Urine pregnancy test is required prior to first administration of study treatment if more than 7 days have elapsed from baseline serum pregnancy test.

If a Central Venous Access Device (CVAD) is required, at least a 2-day interval between placement of a central line and first bevacizumab administration is recommended.

Treatment Phase (pre- and post-operative) Standard Clinical Assessments

* Physical examination (including basic neurologic exam by investigator)
* ECOG performance status (see Appendix 4)
* Vital signs [weight, body temperature, blood pressure, pulse/ heart rate]
* On each (scheduled) visit, patients will be assessed for adverse events (grading by the common terminology criteria for adverse events (CTCAE version 3.0).

Laboratory Assessments

The following laboratory tests are to be done:

* White blood cell count with differentials (lymphocytes, neutrophils), red blood cell count, hemoglobin, hematocrit and platelet count
* Bilirubin (total and direct), ASAT, ALAT, alkaline phosphatase, albumin, LDH
* Serum creatinine
* Glucose
* Electrolytes (sodium, potassium)
* Calcium
* INR (for patients receiving oral anticoagulant treatment)
* CEA, CA 19-9
* Urinalysis: dip stick test for protein is to be performed before each administration of bevacizumab.
* Serum pregnancy tests (if clinically indicated)

Surgery and Control Visits after Surgery

The first control visit should be performed 10 days after surgery and should include the following assessments:

* ECOG performance status
* Vital signs [weight, body temperature, blood pressure, pulse/ heart rate]
* Haematology, Blood chemistry and Coagulation
* Adverse events (grading by the common terminology criteria for adverse events (CTCAE version 3.0) with special regard to wound healing

The second control visit will be performed 21 days after surgery and should include the same assessments as on the first control visit with the addition of:

* Physical examination
* Electrocardiogram (ECG)
* Tumour Assessment

Final Visit End of treatment safety visit to be performed 28 days after the last drug administration.

Follow up Phase and Termination of Study Progression Free Survival Status and Survival status should be assessed every 3 months for a maximum of 2 years.

STUDY MEDICATION

Dose, Schedule and Administration Bevacizumab Bevacizumab will be given at 5 mg/kg on d1 every two weeks, for 5 consecutive cycles. The 6th cycle will be XELOX without Bevacizumab, allowing for a time window between last administration of Bevacizumab and surgery of 5 weeks.

The time window between surgery and re-start of treatment will be at least 4 weeks and wound healing must be completed. Bevacizumab will then be given at 5 mg/kg on d1 every two weeks, for 6 consecutive cycles in combination with XELOX.

Bevacizumab doses will be calculated for each patient in milligrams per kilogram. The patient's actual weight from the screening visit will be the reference weight throughout the study (i.e., patients will receive the same dose at each treatment). Doses of Bevacizumab will be recalculated for patients who experience more than 10% change in body weight from baseline during the treatment period.

All patients will receive an infusion of study drug in a total volume of 100 mL of 0.9% Sodium Chloride Injection, USP. Bevacizumab infusions should not be administered or mixed with dextrose or glucose solutions.

The initial study drug dose will be delivered over 90 minutes as a continuous IV infusion. If the first infusion is tolerated without infusion associated adverse events the second infusion may be delivered over 60 minutes. If the 60 minute infusion is tolerated, all subsequent infusions may be delivered over 30 minutes. If a patient experiences infusion associated adverse events with the 60 minute infusion, all subsequent doses will be given over 90 minutes. If a patient experiences infusion associated adverse events with the 30 minute infusion, all subsequent doses will be given over 60 minutes.

Should extravasation of the study drug infusion occur, the following steps are to be taken:

1. Discontinue the IV.
2. If a significant volume of the study drug infusion remains, restart the IV at a more proximal site in the same limb
3. Treat the infiltration according to institutional guidelines for infiltration of a noncaustic agent.

In the pre-surgery phase, Bevacizumab will be obtained locally by prescription. After surgery, Bevacizumab will be supplied as glass vials with 4-mL fill, containing 100 mg (25 mg/mL) or with 16-mL fill, containing 400 mg (25 mg/mL). Vials contain no preservative and are for single use only.

Oxaliplatin Liquid Oxaliplatin will be given at 85 mg/m2 on d1 every two weeks, for 6 consecutive cycles, before and after surgery.

Liquid Oxaliplatin dose will be calculated using the body surface area (BSA) of the patient (see Appendix 2). The dose of oxaliplatin administered should be as close as possible to the calculated dose.

Liquid Oxaliplatin administration does not require hyperhydration. In the event of extravasation, administration must be discontinued immediately.

For nausea and vomiting, 5-HT3 antagonists with or without dexamethasone are strongly recommended for oxaliplatin-based chemotherapy.

Liquid Oxaliplatin must be infused either by peripheral vein or central venous line over 2 hours. The infusion line must be adequately flushed with 5% dextrose solution (D5W) between oxaliplatin infusion and the administration of any other drug.

Liquid Oxaliplatin (Eloxatin®) will be obtained locally by prescription.

Capecitabine The dose of Capecitabine is 1.500 mg/m2 twice daily from the evening of d1 until the morning of d8, followed by 1 week rest period. One treatment cycle consists of 2 weeks. Capecitabine will be given for 6 consecutive cycles, before and after surgery.

The appropriate daily dose of capecitabine is identified by determination of the Body Surface Area (see Appendix 2 and 3).

Capecitabine is to be administered orally within 30 minutes after the end of a meal (breakfast, dinner). Tablets should be swallowed with approximately 200 mL water (not fruit juices). The first dose of each cycle will be administered as the evening dose on day 1 and the last dose of each cycle is scheduled the morning of day 8, followed by a 7 day rest period.

Capecitabine (Xeloda®) will be obtained locally by prescription.

Study Treatment Duration In the pre-operative treatment phase 6 cycles of XELOX and 5 cycles of Bevacizumab will be administered, resulting in a total treatment duration of 12 weeks.

Surgery will be performed 2 weeks after the last administration of Capecitabine.

Post-operative treatment consists of 6 cycles XELOX + Bevacizumab and will re-start 4-5 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of metastatic CRC including potentially resectable liver metastases, untreated yet with chemotherapy for metastatic disease
* At least one measurable metastatic lesion (as per RECIST criteria)
* Prior adjuvant or neo-adjuvant chemotherapy/radiotherapy allowed
* ECOG performance status 0 or 1
* Signed written informed consent
* life expectancy greater than 3 months
* patients below 18 years of age
* Adequate haematological function: White blood count ≥ 3 x 1000/L with neutrophils ≥ 1.5 x 1000/L, platelet count ≥ 100 x 1000/L, and hemoglobin ≥ 5.6 mmol/L (9g/dL)
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) range, alkaline phosphatase, Aspartate aminotransferase (ASAT) and Alanin aminotransferase (ALAT) ≤ 5 x ULN
* Serum creatinine ≤ 1.25 ULN and/or creatinine clearance ≥ 60 ml/min
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate 1 g of protein/24 hr
* INR ≤ 1.5 and PTT ≤ 1.5 x ULN within 7 days prior to enrolment
* Women of childbearing potential must have a negative serum pregnancy test done 1 week prior to the administration of the study drug. She and her partner should prevent pregnancy (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) up to at least 6 months after last treatment completion or the last drug dose, whatever happens first.
* Patient must be able to comply with the protocol

Exclusion Criteria

* Extrahepatic disease, except concurrent diagnosis of primary CRC
* Prior chemotherapeutic treatment for metastatic CRC
* Serious, non healing wound, ulcer, or bone fracture.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment,
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication
* Pregnancy (absence to be confirmed by ß-HCG test) or lactation
* Men of childbearing potential not willing to use effective means of contraception
* Previous exposure to anti-VEGF antibodies
* Treatment with any investigational agent(s) within 4 weeks prior to study entry
* Known allergic/hypersensitivity reaction to any of the components of study treatments
* Clinically significant cardiovascular disease, for example CVA (6 months before treatment start), myocardial infarction (6 months before treatment start), unstable angina, NYHA grade 2 CHF, or uncontrolled hypertension.
* History of significant neurologic or psychiatric disorders including dementia, seizures, bipolar disorder
* Medical or psychological condition that would not permit the patient to complete the study or sign informed consent
* Known alcohol or drug abuse
* Clinical or radiological evidence of CNS metastases.
* Past or current history (within the last 2 years prior to treatment start) of other malignancies except metastatic colorectal cancer (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
* History of thromboembolic or haemorrhagic events within 6 months prior to treatment.
* Evidence of bleeding diathesis or coagulopathy
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes i.e. except for anticoagulation for maintenance of patency of permanent indwelling IV catheters.
* Chronic daily treatment with aspirin (> 325 mg/day) or clopidogrel (>75 mg/day).
* Chronic daily treatment with corticosteroids (dose of 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
* Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial
* gastrointestinal ulceration
* Known peripheral neuropathy NCI CTC Grade 1. Absence of deep tendon reflexes (DTRs) as the sole neurological abnormality does not render the patient ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is the Resectability (R0) rate after neoadjuvant Bevacizumab in potentially resectable mCRC. | 4 months

SECONDARY OUTCOMES:
Feasibility with regards to GI bleeding and wound healing complications after surgery of liver metastases | 1 month
Overall Response Rate (ORR) | 4 months
Recurrence Free Survival (RFS) | 3 years
Overall Survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gruenberger, MD, Principal Investigator — Austrian Society Of Surgical Oncology
Locations (1):
- Medical University Hospital Vienna, Vienna, Vienna, Austria